CLINICAL TRIAL: NCT01123304
Title: A Phase 1 Clinical Trial of Intra-Tumoral Injection of Human IgM Monoclonal Antibody (MORAb-028) to the Ganglioside GD2 in Subjects With Injectable Metastatic Melanoma
Brief Title: Safety Study of Human IgM (MORAb-028) to Treat Metastatic Melanoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This study has been terminated due to lack of availability of investigational product.
Sponsor: Morphotek (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MORAb028-002
Record Dates: First submitted 2010-05-12; First posted 2010-05-14 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-07

CONDITIONS: Melanoma
Keywords: melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MORAb 028 (Experimental)
  Interventions: Drug: MORAb028

INTERVENTIONS:
Drug: MORAb028 — 1 mg MORAb-028 will be injected at either 1 mg/cm3 per day over 5 days for a total dose of 5 mg for the first cohort and 2 mg/cm3 for the second cohort. Subjects will receive MORAb-028 injections on Days: 1-5, 8-12 and 22-26.

SUMMARY:
This research is being done to find out the safety of MORAb-028 in subjects with metastatic melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed AJCC Stage IIIB, IIIC or IV melanoma with injectable metastases (in transit, intradermal, or subcutaneous nodules)
* Tumor accessible to intra-tumoral injections
* Cumulative tumor volume great enough to accept MORAb-028 injections for a given dose level, based on intent to inject at a concentration of 1 mg/cm3

Exclusion Criteria:

* Are candidates for curative surgical excision or lymphadenectomy
* Prior non-surgical treatment within 4 weeks
* Known central nervous system (CNS) tumor involvement or metastases
* Hypersensitivity to MORAb-028

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-05; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Safety of multiple intralesional administration of MORAb-028 | Day 33
  After each patient completes study treatment the patient is evaluated for dose limiting toxicities (DLTs) up to 1 week after their last dose (at day 33)

SECONDARY OUTCOMES:
Maximum tolerated dose of intralesional administration of MORAb-028 | 22 months

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Wallin, MD, Study Director — Morphotek
Locations (1):
- John Wayne Cancer Institute, Santa Monica, California, United States